CLINICAL TRIAL: NCT04466839
Title: Evaluation of the Containment Impact Linked to the Covid-19 Pandemic in a Population of Parkinson Patients
Acronym: ERCO-Park
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0193
Record Dates: First submitted 2020-06-23; First posted 2020-07-10 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease; COVID
Keywords: Parkinson Disease,; COVID-19; Confinement
MeSH Terms: conditions — Parkinson Disease; COVID-19 | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parkinsonian patients: Cohort of parkinsonian patients followed by doctors from the Parkinson Expert Centers in teaching hospitals.
  Interventions: Other: Questionnaire and interview

INTERVENTIONS:
Other: Questionnaire and interview — The questionnaires are Parkinson Disease Questionnaire-8 Items (PDQ-8) Visual Analog Scale (VAS) is visual analog scale visual numeric from 0 to 100, Neuropsychiatric Inventory-Questionnaire-Reduced (NPI-R) and Clinical Global Impression-Impairment (CGI-I).

SUMMARY:
The consequences of COVID-19 in these already fragile patients should be evaluated. It will be important to appreciate the confinement consequences imposed on the patient on the course and impact of the disease.

These consequences can be assessed by the end of confinement and 6 months after the latter is lifted.

DETAILED DESCRIPTION:
Adaptation capacities are necessary to cope with the brutal and drastic changes imposed by the pandemic and its consequences. In Parkinson's disease, where there are routine situations with difficulties adjusting to newness, patients in the current situation may be particularly affected and present anxiety due to great difficulties in adaptation.

The repercussions in terms of symptoms (motor and non-motor) of the disease could be very significant. In this population already widely exposed to anxio-depressive symptoms (depression being a common symptom of Parkinson's disease, affecting up to 30 to 40% of patients outside of crisis periods), we can expect a risk increased psychiatric decompensation. The psychiatric consequences could not be limited to the current period but also concern long-term patients, in particular if there is decompensation of other symptoms of the disease (motors, complications linked to treatment, etc.).

The consequences of COVID-19 in these already fragile patients should be evaluated. It will be important to appreciate the confinement consequences imposed on the patient on the course and impact of the disease.

These consequences can be assessed by the end of confinement and 6 months after the latter is lifted.

This is an observational, French multicenter study, of an uncontrolled cohort of parkinsonian patients followed by doctors from Parkinson Expert Centers in hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed by a doctor from the Parkinson Expert Center of the Toulouse University Hospital, Lille, Paris, Rouen, Nimes, Reims, Besancon, Marseille
* And with idiopathic Parkinson's disease
* Patients hospitalized or in consultation between 16/03/2020 and 16/05/2020.

Exclusion Criteria:

* Atypical parkinsonian syndrome
* Patient subject to a legal protection order (tutorship)
* Patient not wishing to answer questions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient followed by a doctor from the Parkinson Expert Center with idiopathic Parkinson's disease between 16/03/2020 and 16/05/2020.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Impact of containment related to the Covid-19 pandemic. | 6 months after the end of the pandemic
  To compare quality of life using Parkinson Disease Questionnaire-8 Items (PDQ-8 ), during the period of confinement linked to the Covid-19 pandemic and 6 months after the end of the pandemic in patients with idiopathic Parkinson's disease.
  The minimum value is "never" and maximum value is "always"

SECONDARY OUTCOMES:
Conditions of containment during the Covid-19 pandemic. | Day 1
  Describe in a cohort of Parkinson's patients the conditions of confinement during the confinement period linked to the Covid-19 pandemic such as lifestyle (patient living alone, patient living with a caregiver, patient living in nursing home) and continuing paramedical care (physiotherapist, speech therapist), thanks to a psychosocial assessment
The number of patients infected or possibly infected with Covid-19 | 6 months after the end of the pandemic
  Infected patients will be defined as having had a positive polymerase chain reaction (PCR) or compatible chest scanner. Patients potentially infected: patients who presented symptoms during the period which could suggest an infection by the Covid-19 virus: cough, fever and dyspnea
Symptoms modifications | 6 months after the end of the pandemic
  Patients will be asked to list the 3 main symptoms that have changed during the confinement period

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne ORY MAGNE, Principal Investigator — University Hospital, Toulouse
Locations (8):
- France (8):
  - Centre Hospitalier Régionale Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire Lille, Lille
  - Centre Hospitalier Universitaire de Marseille, Marseille
  - Centre Hospitalier Universitaire de Nîmes - Caremeau, Nîmes
  - Centre Hospitalier Universitaire de la Pitié-Salpêtrière, Paris
  - Centre Hospitalier Universitaire de Reims, Reims
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fabbri M, Leung C, Baille G, Bereau M, Brefel Courbon C, Castelnovo G, Carriere N, Damier P, Defebvre L, Doe de Maindreville A, Fluchere F, Fuzzatti M, Grabli D, Maltete D, Rousseau V, Sommet A A, Thalamas C, Thiriez C, Rascol O, Ory-Magne F. A French survey on the lockdown consequences of COVID-19 pandemic in Parkinson's disease. The ERCOPARK study. Parkinsonism Relat Disord. 2021 Aug;89:128-133. doi: 10.1016/j.parkreldis.2021.07.013. Epub 2021 Jul 13. PMID 34293534